CLINICAL TRIAL: NCT01120548
Title: SLEEP DISORDERED BREATHING DURING CARDIAC REHABILITATION A Study of the Improvement in Physical Performance of Patients With Heart Failure During Cardiac Rehabilitation Due to the Correction of Sleep Disordered Breathing
Brief Title: Sleep Apnea Treatment During Cardiac Rehabilitation of Congestive Heart Failure Patients
Acronym: SATELIT-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: ResMed (Industry); ResMed Foundation (Other); Adep Assistance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-07
Record Dates: First submitted 2010-05-06; First posted 2010-05-11 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure; Sleep Disordered Breathing
Keywords: CARDIAC REHABILITATION; Nocturnal Ventilation; Apnea hypopnea index is > 15/h
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation + Ventilation Group (Experimental): Patient Heart Failure with sleep disordered breathing who follows ventilation therapy and physical training.
  Interventions: Other: ventilation therapy
- Rehabilitation Only Group (No Intervention)

INTERVENTIONS:
Other: ventilation therapy — The service provider will provide the patient with the ventilation device and will explain to the patient how to operate the device and how to fit the mask according to the specifications.
  There will be an oximetry recording during ventilation on the first night. After the first night, the ventilation parameters recorded by the machine and the oximetry results will be read and used to adjust the settings.
  Starting the first week and at the end of the programme, the following ventilation parameters will be collected: compliance, leaks, AHI, ventilation mode, pressures used. The threshold of length of nocturnal ventilation fixed to 3h per night on average in order to consider a compliant patient.
  Arms: Rehabilitation + Ventilation Group

SUMMARY:
Sleep disordered breathing (SDB) is a frequent comorbidity for heart failure patients. Its prevalence varies according to the seriousness of the condition of the patients, but it is present in approximately 50% of patients. Screening patients for SDB and managing them by providing adapted ventilation therapy should improve their quality of life or even their prognosis. Moreover, SDB lowers nocturnal cardiovascular recovery abilities and leads to an increase in fatigability and, as a result, exercise intolerance in patients with heart failure. Physical training as part of a cardiac rehabilitation programme provides many benefits, including improving patients' exercise capacities. Our hypothesis is that adapted sleep disordered breathing therapy during rehabilitation will lead to an improvement in rehabilitation results.

DETAILED DESCRIPTION:
Controlled, randomised, multicentre study. Patients will be assessed prior to starting the rehabilitation programme with regard to exercise tolerance parameters (cardiopulmonary exercise test, 6 minute walk test), ultrasound parameters and biological parameters (Na, Hb, BNP).

The cardiac rehabilitation programme will include education, secondary prevention and physical training components in each of the two groups. The physical training component will include a minimal "base" of activities that is identical for both groups. The nocturnal therapy device will be adapted to the type of SDB specific to each patient (central, mixed, obstructive). The randomisation will be stratified by centre according to predictive factors for performance improvement during rehabilitation.

The main objective is to evaluate the improvement in physical performance resulting from adapted ventilation on SDB compared to physical training alone in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have NYHA class II to IIIb heart failure, operated or not, ischemic or not, without significant valve pathology.
* Referred to cardiac rehabilitation
* With an EF < 40%
* And an apnea-hypopnea index > 15/h (determined by a nasal flow recording method)
* Have signed the consent document to participate in the study.

Exclusion Criteria:

* Patients who have been stabilised for less than 10 days (inotropic drugs or modification of the anticipated resynchronisation or PM parameters)
* Patients who already use sleep disordered breathing devices
* Resting SBP < 80 mmHg (averaged over 3 separate measurements)
* Recent angioplasty (within the last 10 days)
* Infarction within the last 10 days
* Heart surgery within the last 15 days
* Valve dysfunction requiring surgery
* Uncontrolled high blood pressure (BP > 180 and/or 110 mmHg)
* Anaemia (Hb < 9g/dl)
* Haemodialysis
* Patient receiving circulatory assistance
* Severe chronic respiratory failure (FEV1 < 1000) or hypercapnia greater than 46 mmHg
* Patient incapable of performing a 6 minute walk test and an exercise test
* Absolute contraindication for an exercise test and/or physical training according to the recommendations of the French Society of Cardiology
* Evolving myopericarditis
* Severe ventricular rhythm disorders that do not stabilise with treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Peak VO2 | Day 1
  The primary endpoint is the relative improvement of exercise tolerance, estimated using the changes in the patient's peak VO2 measured before starting and after finishing the rehabilitation programme between the both group.
Peak VO2 | Between 4 to 9 weeks
  The primary endpoint is the relative improvement of exercise tolerance, estimated using the changes in the patient's peak VO2 measured before starting and after finishing the rehabilitation programme between the both group.

SECONDARY OUTCOMES:
Physical training compliance | between 4 and 9 weeks
  Secondary endpoints include compliance with rehabilitation sessions, estimated by comparing the number of sessions in which training was effectively carried out with the anticipated number of sessions and other exercise tolerance parameters (maximum power, duration of exercise, submaximal parameters) in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Corone, MD, Principal Investigator — Centre Médical de Bligny; Marie-Christine Iliou, MD, Principal Investigator — Hôpital Corentin Celton
Locations (19):
- France (19):
  - Centre Médical de Bligny, Briis-sous-Forges
  - Clinique de Châtillon, Châtillon
  - Hôpital Albert Chenevier, Créteil
  - Dieulefit Santé, Dieulefit
  - Hôpital Arthur Gardiner, Dinard
  - Clinique de cardiopneumologie, Durtol
  - Hôpital Sud - Institut de Rééducation, Échirolles
  - Hôpital Corentin Celton, Issy-les-Moulineaux
  - Clinique de La Mitterie, Lomme
  - Centre IRIS, Marcy-l'Étoile
  - Centre Cardio-Vasculaire Valmante, Marseille
  - Clinique de réadaptation cardiaque Cardiocéan, Puilboreau
  - Hôpital Nord 6, Saint-Etienne
  - Hôpital Intercommunal Sud Léman Valserine, Saint-Julien-en-Genevois
  - Centre William Harvey - le Haut Boscq, Saint-Martin-d'Aubigny
  - Centre de réadaptation cardiaque Leopold Bellan, Tracy-le-Mont
  - Institut Régional de Réadaptation, Vandœuvre-lès-Nancy
  - La Maison du Mineur, Vence
  - Centre Hospitalier Calmette, Yerres